CLINICAL TRIAL: NCT04462003
Title: Efficacy and Safety of Apixaban in Patients With Active Malignancy and Acute Deep Venous Thrombosis.
Brief Title: Efficacy of Apixaban in Malignancy With Deep Venous Thrombosis
Acronym: DVT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mostafa El Mokadem, Dr, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Apixaban in DVT with cancer
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Deep Vein Thrombosis; Malignancy
MeSH Terms: conditions — Venous Thrombosis; Neoplasms | interventions — apixaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apixaban (Active Comparator): 50 patients with DVT with malignancy were randomized to apixaban 10 mg twice daily dose for 7 days followed by apixaban 5 mg twice daily
  Interventions: Drug: Apixaban
- Enoxaparin (Active Comparator): 50 patients with DVT with malignancy were randomized to enoxaparin (1mg/Kg/SC every 12 h)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Apixaban — 10 mg/12 h for 1 week followed by 5 mg/12 h
  Arms: Apixaban
Drug: Enoxaparin — 1mg/Kg/sc/12h
  Arms: Enoxaparin

SUMMARY:
The aim of study was to evaluate the efficacy and safety of Apixaban in patients with acute deep venous thrombosis and active malignancy compared with weight adjusted subcutaneous (LMWH). It was hypothesised that Apixaban could be as effective as rivaroxiban and edoxaban in treatment of patients with acute DVT and active malignancy with a lower risk of bleeding especially in those with GIT cancer.

DETAILED DESCRIPTION:
Patients with active malignancy have hypercoagulable state particularly, those receiving intravenous chemotherapy, with six fold higher risk of venous thromboembolism (VTE) [1]. Anticoagulation for malignancy associated deep venous thrombosis (DVT) can be difficult because of different limitations like bleeding, drug-drug interactions with chemotherapy and inconvenience with repeated subcutaneous injections of low-molecular-weight heparin (LMWH) [2]. In comparison with patients without active malignancy, patients with cancer who are on warfarin therapy have 2 to 6 folds more major bleeding events and 2 to 3 times more VTE recurrence [3,4]. The American College of Chest Physicians Guidelines recommended (LMWH) as standard therapy for management of acute VTE in patients with active malignancy [5]. Recently, Rivaroxiban and Edoxaban were considered as an alternative to weight-adjusted subcutaneous LMWH after pulmonary embolism in patients with active cancer without gastrointestinal (GIT) malignancy [6]. Apixaban is a direct factor Xa inhibitor approved by FDA for treatment of DVT and VTE [7]. However its efficacy in management of acute DVT and VTE associated with cancer is still unresolved issue. The aim of study was to evaluate the efficacy and safety of Apixaban in patients with acute deep venous thrombosis and active malignancy compared with weight adjusted subcutaneous (LMWH).

ELIGIBILITY:
Inclusion Criteria Patients with active malignancy presenting with acute deep venous thrombosis and still treated with chemotherapy

Exclusion Criteria:

* Patients with pulmonary embolism and hemodynamic instability requiring thrombolytic therapy
* Previous DVT or venous thromboembolism
* Administration of LMWH or unfractionated heparin before randomization
* Brain tumours, cerebral metastes, hepatic tumours or impairment Child-Pugh B or C, -Recent or current active or life threating bleeding (e.g. intr acranial haemorrhage or gastrointestinal bleeding)
* Thrombocytopenia (platelets <100 x 109L)
* Severe chronic kidney disease (estimated glomerular filtration rate <30 ml/minute)
* Pregnant women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-07-02 (Estimated); Study Completion 2020-07-03 (Estimated)

PRIMARY OUTCOMES:
Recurrent deep venous thrombosis or venous thromboembolism | 6 months
  New or non resolving completely occluded deep venous thrombosis or occurrence of pulmonary embolism
Occurrence of fatal or major bleeding | 6 months
  Need for hospitalization, blood transfusion, surgical intervention or resulting into death
Mortality related to massive pulmonary embolism | 6 months
  Death caused by hemodynamic instability secondary to massive pulmonary embolism

SECONDARY OUTCOMES:
Occurrence of non-fatal or minor bleeding | 6 months
  Bleeding that does not need hospitalization, blood transfusion, surgical intervention or resulting into death

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa E Mokadem, Principal Investigator — Faculty of Medicine, Beni-Suef University
Locations (1):
- Faculty of Medicine,Beni-Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med. 2000 Mar 27;160(6):809-15. doi: 10.1001/archinte.160.6.809. PMID 10737280
- [Result] Ay C, Beyer-Westendorf J, Pabinger I. Treatment of cancer-associated venous thromboembolism in the age of direct oral anticoagulants. Ann Oncol. 2019 Jun 1;30(6):897-907. doi: 10.1093/annonc/mdz111. PMID 30918939
- [Result] Hutten BA, Prins MH, Gent M, Ginsberg J, Tijssen JG, Buller HR. Incidence of recurrent thromboembolic and bleeding complications among patients with venous thromboembolism in relation to both malignancy and achieved international normalized ratio: a retrospective analysis. J Clin Oncol. 2000 Sep;18(17):3078-83. doi: 10.1200/JCO.2000.18.17.3078. PMID 10963635
- [Result] Prandoni P, Lensing AW, Piccioli A, Bernardi E, Simioni P, Girolami B, Marchiori A, Sabbion P, Prins MH, Noventa F, Girolami A. Recurrent venous thromboembolism and bleeding complications during anticoagulant treatment in patients with cancer and venous thrombosis. Blood. 2002 Nov 15;100(10):3484-8. doi: 10.1182/blood-2002-01-0108. Epub 2002 Jul 12. PMID 12393647
- [Result] Kearon C, Akl EA, Ornelas J, Blaivas A, Jimenez D, Bounameaux H, Huisman M, King CS, Morris TA, Sood N, Stevens SM, Vintch JRE, Wells P, Woller SC, Moores L. Antithrombotic Therapy for VTE Disease: CHEST Guideline and Expert Panel Report. Chest. 2016 Feb;149(2):315-352. doi: 10.1016/j.chest.2015.11.026. Epub 2016 Jan 7. PMID 26867832
- [Result] Konstantinides SV, Meyer G, Becattini C, Bueno H, Geersing GJ, Harjola VP, Huisman MV, Humbert M, Jennings CS, Jimenez D, Kucher N, Lang IM, Lankeit M, Lorusso R, Mazzolai L, Meneveau N, Ni Ainle F, Prandoni P, Pruszczyk P, Righini M, Torbicki A, Van Belle E, Zamorano JL; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of acute pulmonary embolism developed in collaboration with the European Respiratory Society (ERS). Eur Heart J. 2020 Jan 21;41(4):543-603. doi: 10.1093/eurheartj/ehz405. No abstract available. PMID 31504429
- [Result] Agnelli G, Buller HR, Cohen A, Gallus AS, Lee TC, Pak R, Raskob GE, Weitz JI, Yamabe T. Oral apixaban for the treatment of venous thromboembolism in cancer patients: results from the AMPLIFY trial. J Thromb Haemost. 2015 Dec;13(12):2187-91. doi: 10.1111/jth.13153. Epub 2015 Oct 29. PMID 26407753
- [Result] McBane RD 2nd, Wysokinski WE, Le-Rademacher JG, Zemla T, Ashrani A, Tafur A, Perepu U, Anderson D, Gundabolu K, Kuzma C, Perez Botero J, Leon Ferre RA, Henkin S, Lenz CJ, Houghton DE, Vishnu P, Loprinzi CL. Apixaban and dalteparin in active malignancy-associated venous thromboembolism: The ADAM VTE trial. J Thromb Haemost. 2020 Feb;18(2):411-421. doi: 10.1111/jth.14662. Epub 2019 Nov 28. PMID 31630479
- [Result] Agnelli G, Becattini C, Bauersachs R, Brenner B, Campanini M, Cohen A, Connors JM, Fontanella A, Gussoni G, Huisman MV, Lambert C, Meyer G, Munoz A, Abreu de Sousa J, Torbicki A, Verso M, Vescovo G; Caravaggio Study Investigators. Apixaban versus Dalteparin for the Treatment of Acute Venous Thromboembolism in Patients with Cancer: The Caravaggio Study. Thromb Haemost. 2018 Sep;118(9):1668-1678. doi: 10.1055/s-0038-1668523. Epub 2018 Aug 13. PMID 30103252
- [Result] Cheung KS, Leung WK. Gastrointestinal bleeding in patients on novel oral anticoagulants: Risk, prevention and management. World J Gastroenterol. 2017 Mar 21;23(11):1954-1963. doi: 10.3748/wjg.v23.i11.1954. PMID 28373761
- [Result] Desai J, Kolb JM, Weitz JI, Aisenberg J. Gastrointestinal bleeding with the new oral anticoagulants--defining the issues and the management strategies. Thromb Haemost. 2013 Aug;110(2):205-12. doi: 10.1160/TH13-02-0150. Epub 2013 May 23. No abstract available. PMID 23702623
- [Result] Desai J, Granger CB, Weitz JI, Aisenberg J. Novel oral anticoagulants in gastroenterology practice. Gastrointest Endosc. 2013 Aug;78(2):227-39. doi: 10.1016/j.gie.2013.04.179. Epub 2013 May 29. No abstract available. PMID 23725876
- [Result] Cannon CP, Kohli P. Danger ahead: watch out for indirect comparisons! J Am Coll Cardiol. 2012 Aug 21;60(8):747-8. doi: 10.1016/j.jacc.2012.05.012. No abstract available. PMID 22898071
- [Derived] Mokadem ME, Hassan A, Algaby AZ. Efficacy and safety of apixaban in patients with active malignancy and acute deep venous thrombosis. Vascular. 2021 Oct;29(5):745-750. doi: 10.1177/1708538120971148. Epub 2020 Nov 5. PMID 33153401